CLINICAL TRIAL: NCT07113132
Title: Role of SF3B1 Mutation in Assessment of Acute and Chronic Lymphatic Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Safaa Ali (Other)
Responsible Party: Sponsor-Investigator, Safaa Ali, assisstant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: sf3b1 mutation in ALL and CLL
Record Dates: First submitted 2025-07-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia ALL; Chronic Lymphocytic Leukemia (CLL)
Keywords: sf3b1 mutation; all; cll
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — peripheral blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- all patients group: peripheral blood samples of 28 acute lymphoblastic leukemia patients
- cll patients: peripheral blood samples of 28 chronic lymphocytic leukemia patients
- control group: peripheral blood samples of 28 control

SUMMARY:
aim of the work

1. To evaluate the presence of SF3B1-K700E mutation in acute lymphoblastic leukemia and chronic lymphocytic leukemia.
2. To determine the correlation between the presence of SF3B1-K700E mutation with other laboratory findings.

DETAILED DESCRIPTION:
Leukemia is one of the deadliest diseases having negative impact on people all over the world. Acute Lymphocytic Leukemia (ALL) is a type of WBC cancer, it's a rapidly invasive disease that originates from B- or T-lymphocyte progenitors. Accumulation of lymphoblasts and suppression of normal cells are the main characteristics of the disease course .

Acute lymphoblastic leukemia (ALL) predominantly affects children, with an incidence of 3-4/100,000 in patients under 14 years of age. The five-year survival rate is approximately 90% in children and 65% in adults .

The French-American-British (FAB) categorizes ALL into three subtypes However, the WHO classification incorporates immunophenotypic and genetic details, offering a more accurate and clinically significant classification, helping to choose therapies and prognostic evaluations according to the distinct characteristics of leukemia. Medical professionals have recently recommended that WHO categorization is better compared to FAB .

Chronic lymphoproliferative diseases (CLPD) are considered as a heterogeneous group of diseases characterized by monoclonal expansion and accumulation of apparently mature lymphocytes, which have a proliferative and/or survival advantage over normal lymphocytes in different organs such as bone marrow, peripheral blood and lymph nodes. This translates into the progressive accumulation of clonal cells and their products, causing peripheral blood and bone marrow lymphocytosis, in addition to lymphadenopathy, splenomegaly or other organomegaly .

Recently, mutations in the genes involved in the spliceosome have attracted considerable interest in different neoplasms. Among the spliceosome mutations, those in the SF3B1 gene are the most frequent and relevant in haematological diseases. Most human genes encode several mRNA isoforms by the alternative splicing process. Because alternatively spliced mRNA isoforms are often associated with cancer, spliceosome mutations have recently sparked significant interest in different neoplasms .

splicing of RNA is a fundamental process in eukaryotes, The spliceosome dynamically assembles on messenger RNA precursors (pre-mRNA), removing introns (regions that do not encode proteins) from pre-mRNA, leaving exons (the remainder of RNA transcription) attached .

It is known that SF3B1 mutations could play multiple roles in the pathogenesis of tumours by dysregulating several cellular functions and pathways, including heme biosynthesis, mitochondrial metabolism, and the NF-κB pathway .

The messenger RNA (mRNA) spliceosome is composed of a complex of five small nuclear ribonucleoproteins (snRNP) U1, U2, U4, U5, and U6 and other proteins and plays critical roles in regulating mRNA splicing and subsequent protein expression. It is assembled through binding of U1 snRNP to the 5' splice site of the pre-mRNA, recruitment of U2snRNP to the 3' splicing site at the intron-exon junction guided by the branch region sequence, and joining of the tri-snRNP U4/U5/U6 .

SF3B1, an essential protein in the U2snRNP complex, facilitates U2snRNP binding at the branch point near the 3' splicing site. SF3B1 mutants were shown to alter U2snRNP function by promoting alternative branch-point usage and induction of cryptic 3' splice site selection, thereby generating aberrantly spliced mRNA transcripts subject to nonsense-mediated decay and downregulation of target transcripts and protein expression .

The SF3B1 gene is located on the long arm of chromosome 2 (2q33.1) and encodes for the biggest subunit (155 KDa) of the splicing factor 3b protein complex . The interaction between the SF3B1 complex, the 12S unit, and the splicing factor 3a complex gives rise to the U2 small nuclear ribonucleoproteins (snRNP), fundamental for spliceosome assembly and mRNA splicing . The SF3B1 protein is located principally in the nucleus, where it forms nuclear speckles; it is necessary to anchor U2 snRNP to the pre-mRNA by sequence-independently binding the intron branch site .

SF3B1 high proportion in hematopoietic malignancies occurs within codon 700 (K700E) located in the HEAT domain repeat sequence. In addition, hotspots such as R625, K666, and H662 also occur in some proportion , which are thought to have similar mutational functions due to their spatial proximity to K700E in HEAT repeats. .

The most common SF3B1 mutation is an A to G transition that results in lysine to glutamic acid substitution at amino acid position 700 (SF3B1-K700E) .

Mutated SF3B1 gives rise to a protein with a neomorphic activity linked to several mechanisms involved in RNA processing. About half of aberrantly spliced mRNAs are characterized by the presence of premature stop codons, resulting in nonsense-mediated RNA decay and downregulation of the protein expression. Although the wild-type allele is still able to be expressed, the amount of protein produced is unable to compensate for the mutant allele. Another possibility is the translation of new proteins that lack the correct biological function and/or that acquire aberrant functions .

A study has shown Hotspot K700E and non-K700E SF3B1mut MDS show distinct clinical and mutational profiles in MDS, with K700E showing significantly better Overall survival than non-K700E and SF3B1wt. Only the absence of the SF3B1mut K700E mutation independently predicted worse Overall survival in MDS. Hence, identification of the SF3B1 mutation type is important for risk stratification .

In the study by Wang and colleges, somatic mutations of SF3B1 were found in approximately 15% of patients, making this the second most frequently mutated gene in CLL .

In a cohort of 537 unselected CLL cases, SF3B1 mutations were present in (8.9%) of cases , The residues surrounding Lys700 were the most frequently mutated (48%) .

Quesada and colleges in 2012 studied 279 untreated patients with CLL and found SF3B1 mutations in 27 (10%) . the most frequent mutation was K700E, occurring in almost half of the cases, No SF3B1 mutation was detected in 156 patients with non-Hodgkin lymphoma . CLL patients with mutations in SF3B1 had more aggressive disease and shorter overall survival than patients without these mutations .

Another study provided evidence that the SF3B1 inhibitor H3B-8800 displays therapeutic effects in mouse models of CLL, particularly when used on CLL cells harbouring SF3B1 mutations .

To address the functional role of SF3B1 in T-ALL, SF3B1 was silenced in T-ALL cell lines using short hairpin RNAs (shRNAs). The cell proliferation rate was significantly decreased upon SF3B1 silencing, accompanied by an increase in apoptotic cell death and G2-M cell cycle arrest. To further assess the role of SF3B1 in disease progression in vivo, SF3B1 was silenced in luciferase-expressing CUTLL1 cells and transplanted the cells into immunocompromised mice. SF3B1 silencing led to a significantly reduced tumour burden and prolonged mouse survival .

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphocytic leukemia or chronic lymphocytic leukemia of both genders at any age.

Exclusion Criteria:

* Patients with any other type of malignancies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study will be conducted on peripheral blood samples of 28 acute lymphoblastic leukemia patients, 28 chronic lymphocytic leukemia patients and 28 control.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
1- To evaluate the presence of SF3B1-K700E mutation in acute lymphoblastic leukemia and chronic lymphocytic leukemia using PCR technique | 2 years
  ARMS PCR technique will be used to detect the presence of SF3B1-MUTATION in acute lymphoblastic leukemia and chronic lymphocytic leukemia
2-To determine the effect of presence of SF3B1-K700E mutation with other laboratory findings. | two years
  determine if the presence of SF3B1-mutation can affect the clinical data as severity of disease or organomegaly and laboratory data as count of white blood cells and platalet and hemoglobin level using automated cbc analyser and bone marrow of the patients (cellularity and count of blast cells) and result of flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Sohair m Farghaly, professor, Study Director — Assiut University; Taghred m Kamal El-Din, asst. prof, Study Chair — Assiut University; Hebatallah Abdellatif, asst. prof, Study Chair — Assiut University; safaa a omran, asst. lect., Principal Investigator — Assiut University

REFERENCES:
- [Background] Cilloni D, Itri F, Bonuomo V, Petiti J. SF3B1 Mutations in Hematological Malignancies. Cancers (Basel). 2022 Oct 8;14(19):4927. doi: 10.3390/cancers14194927. PMID 36230848
- [Background] Wang L, Lawrence MS, Wan Y, Stojanov P, Sougnez C, Stevenson K, Werner L, Sivachenko A, DeLuca DS, Zhang L, Zhang W, Vartanov AR, Fernandes SM, Goldstein NR, Folco EG, Cibulskis K, Tesar B, Sievers QL, Shefler E, Gabriel S, Hacohen N, Reed R, Meyerson M, Golub TR, Lander ES, Neuberg D, Brown JR, Getz G, Wu CJ. SF3B1 and other novel cancer genes in chronic lymphocytic leukemia. N Engl J Med. 2011 Dec 29;365(26):2497-506. doi: 10.1056/NEJMoa1109016. Epub 2011 Dec 12. PMID 22150006
- [Background] Han C, Khodadadi-Jamayran A, Lorch AH, Jin Q, Serafin V, Zhu P, Politanska Y, Sun L, Gutierrez-Diaz BT, Pryzhkova MV, Abdala-Valencia H, Bartom ET, Buldini B, Basso G, Velu SE, Sarma K, Mattamana BB, Cho BK, Obeng RC, Goo YA, Jordan PW, Tsirigos A, Zhou Y, Ntziachristos P. SF3B1 homeostasis is critical for survival and therapeutic response in T cell leukemia. Sci Adv. 2022 Jan 21;8(3):eabj8357. doi: 10.1126/sciadv.abj8357. Epub 2022 Jan 21. PMID 35061527

DOCUMENTS (1):
  • Study Protocol (2025-06-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT07113132/Prot_000.pdf